CLINICAL TRIAL: NCT00848055
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Single Rising, Open-label Doses of AbGn-168 Administered by Intravenous Infusion (1 Mcg/kg, 5 Mcg/kg, 25 Mcg/kg, 125 Mcg/kg, 625 Mcg/kg, 3 mg/kg, or 10 mg/kg) or Subcutaneous Injection (625 Mcg/kg) to Patients With Chronic Plaque Psoriasis
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of AbGn-168 in Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 1240.1
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

ARMS (8):
- arm 1 (Experimental): AbGn168 cohort 1
  Interventions: Drug: AbGn168 intravenous infusion
- arm 2 (Experimental): AbGn168 cohort 2
  Interventions: Drug: AbGn168 intravenous infusion
- arm 3 (Experimental): AbGn168 cohort 3
  Interventions: Drug: AbGn168 intravenous infusion
- arm 4 (Experimental): AbGn168 cohort 4
  Interventions: Drug: AbGn168 intravenous infusion
- arm 5 (Experimental): AbGn168 cohort 5
  Interventions: Drug: AbGn168 intravenous infusion
- arm 6 (Experimental): AbGn168 cohort 6
  Interventions: Drug: AbGn168 intravenous infusion
- arm 7 (Experimental): AbGn168 cohort 7
  Interventions: Drug: AbGn168 intravenous infusion
- arm 8 (Experimental): AbGn168 cohort 8
  Interventions: Drug: AbGn168 subcutaneous injection

INTERVENTIONS:
Drug: AbGn168 intravenous infusion — single dose intravenous infusion
  Arms: arm 2
Drug: AbGn168 intravenous infusion — single dose intravenous infusion
  Arms: arm 3
Drug: AbGn168 intravenous infusion — single dose intravenous infusion
  Arms: arm 1
Drug: AbGn168 intravenous infusion — single dose intravenous infusion
  Arms: arm 4
Drug: AbGn168 intravenous infusion — single dose intravenous infusion
  Arms: arm 5
Drug: AbGn168 intravenous infusion — single dose intravenous infusion
  Arms: arm 6
Drug: AbGn168 intravenous infusion — single dose intravenous infusion
  Arms: arm 7
Drug: AbGn168 subcutaneous injection — single dose subcutaneous injection
  Arms: arm 8

SUMMARY:
The general aim of the trial is to determine the safety, tolerability and pharmacologic profile of single escalating doses of AbGn-168 administered subcutaneously or intravenously to patients with chronic plaque psoriasis

ELIGIBILITY:
Inclusion criteria:

Patients with chronic plaque psoriasis covering at least 3% of body surface area. Female subjects must be postmenopausal or surgically sterilized.

Exclusion criteria:

Recent use of biologic agents, oral psoriasis medications or phototherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety measurements including physical examination, vital signs, ECG, clinical laboratory tests, and adverse events | Baseline, on treatment,and at end of study

SECONDARY OUTCOMES:
Pharmacokinetic and pharmacodynamic endpoints including Cmax, tmax, AUC, t1/2, CL and Vss, target lesion assessment and skin biopsy | Baseline and on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- United States (6):
  - 1240.1.05 Boehringer Ingelheim Investigational Site, Boise, Idaho
  - 1240.1.06 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1240.1.04 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1240.1.02 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1240.1.01 Boehringer Ingelheim Investigational Site, New York, New York
  - 1240.1.03 Boehringer Ingelheim Investigational Site, Dallas, Texas
- 1240.1.7 Boehringer Ingelheim Investigational Site, Berlin, Germany